CLINICAL TRIAL: NCT00556738
Title: Intrapulmonary Percussive Ventilation and Nasal Continuous Positive Airway Pressure Ventilation in Transient Respiratory Distress of the Newborn: A Randomized Controlled Trial
Brief Title: Intrapulmonary Percussive Ventilation (IPV) Versus Nasal Continuous Positive Airway Pressure Ventilation (nCPAP) in Transient Respiratory Distress of the Newborn
Acronym: HFPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical research and Innovation director, University hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2007/09; 2007-A00666-47
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: HFPV; neonatal respiratory distress
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Pulmonary Atelectasis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nHFPV (Experimental): Intrapulmonary Percussive Ventilation
  Interventions: Procedure: Intrapulmonary Percussive Ventilation
- nCPAP (Active Comparator): Nasal Continuous Positive Airway Pressure ventilation
  Interventions: Procedure: Nasal Continuous Positive Airway Pressure ventilation

INTERVENTIONS:
Procedure: Nasal Continuous Positive Airway Pressure ventilation — Nasal Continuous Positive Airway Pressure ventilation
  Arms: nCPAP
Procedure: Intrapulmonary Percussive Ventilation — Intrapulmonary Percussive Ventilation
  Arms: nHFPV

SUMMARY:
During caesarean section, transient respiratory distress which occurs frequently (3%) with possible complications are at present managed by non invasive nasal continuous positive airway pressure ventilation (nCPAP) associated with oxygen therapy. Intrapulmonary Percussive Ventilation (IPV) is a non-invasive ventilatory mode used in some intensive care units to treat some respiratory distress syndrome of the newborn with a good tolerance, but without evaluation in prospective studies

DETAILED DESCRIPTION:
* Principal Objective: To show that IPV ventilation can decrease the duration of transient respiratory distress as well as the risk of complications.
* Secondary Objective: Comparison between the two groups regarding: Length of oxygen therapy, complications (pneumothorax, pulmonary infections), need for intensive care hospitalization
* Study design: Open, prospective randomized trial.
* Inclusion criteria: Neonates with gestational age ≥ 35 weeks and weight ≥ 2000g, caesarean section, respiratory distress syndrome (modified Silverman score > 5, SpO2 < 90%), management within 20 minutes after birth.
* Exclusion criteria: clinical thoracic retraction, congenital lung malformation, meconium aspiration, neonatal infection, other congenital malformations.
* Study plan: After the screening evaluation and written consent document, neonates will be randomized into two groups: nCPAP ventilation or IPV. During the 6 hours after randomization, clinical data will be monitored: cardiac and respiratory frequency (CF -RF), saturation (SaO2), oxygenotherapy, Silverman Score. Then, neonates will be supervised 3 days after normalization of the respiratory distress.
* Number of subjects: 100 (50 in each group)

ELIGIBILITY:
Inclusion Criteria:

* Caesarean newborn
* Gestational age ≥ 35 weeks
* Weight ≥ 2 kg
* SaO2 < 90% after 10 min of life
* Silverman score ≥ 5
* Treated less than 20 min after birth
* Social security affiliation (parents)
* Informed consent signed (parents)

Exclusion Criteria:

* Thoracic retraction
* Congenital intrathoracic malformations
* Meconium aspiration
* Early neonatal infections with hemodynamic troubles
* Severe neonatal asphyxia
* Polymalformative syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Difference in time (min) required to normalize the respiratory distress (modified Silverman score = 0, no need for oxygen, RF < 50 bpm and SaO2 > 92%) between the two ventilatory modes | Within the first 6 hours after birth

SECONDARY OUTCOMES:
Number of pneumothorax, lung infections, transfer to intensive care service, time of oxygenotherapy | Within the first 72 hours after birth

CONTACTS AND LOCATIONS:
Overall Officials: Clothilde Bertrand, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Néonatalogie - Maternité - Hôpital Pellegrin, Bordeaux, France

REFERENCES:
- [Derived] Dumas De La Roque E, Bertrand C, Tandonnet O, Rebola M, Roquand E, Renesme L, Elleau C. Nasal high frequency percussive ventilation versus nasal continuous positive airway pressure in transient tachypnea of the newborn: a pilot randomized controlled trial (NCT00556738). Pediatr Pulmonol. 2011 Mar;46(3):218-23. doi: 10.1002/ppul.21354. Epub 2010 Oct 20. PMID 20963833